CLINICAL TRIAL: NCT01385332
Title: A Comparative Study of Two Patterns of Controlled Ovarian Hyperstimulation in Mid Follicular Phase or Early Luteal Phase for Egg Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Miguel Angel Checa, MD, Parc de Salut Mar
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UREP-ONCO-2010
Record Dates: First submitted 2010-05-28; First posted 2011-06-30 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Stimulation in the Ovary
Keywords: Metaphase II; Ovarian stimulation; Egg donors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early luteal phase -COH- (Active Comparator): We perform an standard antagonist protocol beginning the second day of the menstrual cycle compared with an antagonist protocol beginning in the early luteal phase.
  Interventions: Procedure: Early luteal phase
- Late folicular phase - COH - (Active Comparator): We perform an standard antagonist protocol beginning the second day of the menstrual cycle compared with an antagonist protocol beginning in the late follicular phase.
  Interventions: Procedure: Late follicular phase -COH-

INTERVENTIONS:
Procedure: Early luteal phase — We will administer in the tenth day of the cycle 0.25mg/day of ganirelix until the estradiol levels will be less than 60pgr/mL. Then, we'll start a standard protocol of controlled ovarian hyperstimulation beginning with 150 UI/day. At 6th day of stimulation we'll begin with the antagonist.
  Arms: Early luteal phase -COH-
Procedure: Late follicular phase -COH- — We will administer in the 20th day of the cycle 0.25mg/day of ganirelix until the estradiol levels will be less than 60pgr/mL. Then, we'll start a standard protocol of controlled ovarian hyperstimulation beginning with 150 UI/day. At 6th day of stimulation we'll begin with the antagonist.
  Arms: Late folicular phase - COH -

SUMMARY:
The purpose of this study is to determine the efficacy and safety of two new patterns of controlled ovarian hyperstimulation (defined as total number of picked up eggs). This study will be performed in egg donors but these new patterns will be implemented in fertility preservation patients.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women 18-30 years old, with FSH levels < 10mIU
* irregular menstrual cycle
* BMI between 12-28
* signed inform consent

Exclusion Criteria:

* Polycystic ovarian syndrome, gonadotropins allergy

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of eggs | Participants will be followed after 1-3 hrs of follicular aspiration.
  The results will be presented in one year, egg recipients will be followed until 12 weeks of pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Servei de Ginecologia i Obstetricia, Hospital del Mar-Parc Salut Mar, Barcelona, Spain